CLINICAL TRIAL: NCT03889041
Title: Concerns of Caregivers of Children With Repaired Esophageal Atresia-tracheoesophageal Fistula
Brief Title: Caregivers of Children With Repaired Esophageal Atresia-tracheoesophageal Fistula
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: Dysphagia in esophagealatresia
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Dysphagia; Quality of Life
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers of children with EA-TEF: Caregivers of children with esophageal atresia and tracheoesophageal fistula will be included in the study.
  Interventions: Other: Quality of life assessment

INTERVENTIONS:
Other: Quality of life assessment — The Turkish Feeding/Swallowing Impact Survey will be completed by the caregivers

SUMMARY:
Children with esophageal atresia and tracheoesophageal fistula (EA-TEF) may experience feeding and swallowing difficulties, which result in stressful interactions between children and caregivers, and potentially impact the concerns of caregivers. The aim of this study was to assess concerns of caregivers of children with EA-TEF related to feeding-swallowing difficulties.

DETAILED DESCRIPTION:
Children with repaired esophageal atresia-tracheoesophageal fistula (EA-TEF) experience some degrees of feeding and swallowing difficulties Feeding and swallowing difficulties cause aspiration-induced recurrent pneumonia, malnutrition, dehydration and stressful interactions with their caregivers. There is lack of knowledge regarding the concerns of caregivers of children with EA-TEF related to feeding and swallowing disorders.Therefore, the aim of this study was to assess concerns of caregivers of children with EA-TEF related to feeding-swallowing difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with EA-TEF
* Having a child with swallowing disorders aged between 6 months-18 years

Exclusion Criteria:

* Having a child without swallowing disorders

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Caregivers of children with EA-TEF
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
The Turkish Feeding/Swallowing Impact Survey | 1 month
  The Turkish Feeding/Swallowing Impact Survey (T-FS-IS) is used to describe the quality of life related to activities of daily living, worry and feeding difficulty of caregivers of children. It has 18 questions. Daily activities indicate caregivers' perceptions of time demands on daily activities. Worry is the worry of the caregivers about the children's well-being. Feeding difficulty is related to the challenges during delivery of care specific to feeding/swallowing. Each question of the instrument will be answered on a 5-point Likert scale between 1 to 5. A score of '1' indicates never, and a score of '5' indicates almost always. All scores from 18 questions in the T-FS-IS will be summed, and then divided by 18 to calculate an average total score. Scores within each subscale will also be added together, and then divided by the total number of questions in the subscale to calculate an average subscale score. Higher scores from the instrument represent decreased quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN S ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No